CLINICAL TRIAL: NCT04395846
Title: Heart Failure and Preserved Ejection Fraction: Observation of Its Progression and Prognosis (HOPP-BERN)
Acronym: HOPP-BERN
Status: Active, not recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: HOPP-BERN ( 4236 ); 2019-02018 (Other: BASEC ID 2019-02018)
Record Dates: First submitted 2020-03-25; First posted 2020-05-20 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: CMR; HFpEF; Extracellular Volume; Myocardial Oxygenation; Feature Tracking CMR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Analysis of longitudinal data, cardiovascular magnetic resonance (CMR) imaging and health related data, of patients with heart failure and preserved ejection fraction (HFpEF) over a timeframe of 5 years per patient.

In this study routine clinical data are collected along with additional research parameters measured during CMR. CMR will occur throughout a 5-year follow-up.

DETAILED DESCRIPTION:
Heart Failure with Preserved Ejection Fraction (HFpEF) is becoming increasingly prevalent, yet diagnostics, characterization and prognosis of the disease is still uncertain. Multiple contributing factors have been implicated in the development of HFpEF such as but not limited to myocardial fibrosis, myocardial edema, ventricular remodeling, metabolic dysfunction, coronary microvascular dysfunction, ischemia, systemic effects and associated ventricular-arterial coupling. However, how the longitudinal progression of these factors is associated with HFpEF and whether a causal effect between the pathologic features in HFpEF exist, is not fully understood.

Using cardiovascular magnetic resonance (CMR), multiple cardiac and extracardiac parameters can be investigated in a single non-invasive imaging exam. This will be a single-centre prospective observational longitudinal study with the formation of a database. Patients will undergo a comprehensive CMR exam upon recruitment, 1- and 5-years after enrolment, and also if re-hospitalisation for heart failure occurs. This exam will investigate multiple measures of cardiovascular function, myocardial deformation, edema, fibrosis and oxygenation, 4D haemodynamical assessments, along with measurements of the aorta, liver and spleen. Furthermore, clinical data will be collected for the patients for the creation of a HFpEF database (ie. patient characteristics, Kansas City Cardiomyopathy Questionnaire (KCCQ), HF and risk scores, laboratory biomarkers, diagnostic results). With this study, the investigator will be able to quantify longitudinal changes in CMR features within the HFpEF population, and investigate what features are associated with poor prognosis. The data collected will lead to a greater understanding of HFpEF, and hopefully show which clinical or imaging features can be used to identify, and better risk stratify this heterogenous population.

ELIGIBILITY:
Inclusion Criteria:

* Known Heart Failure with Preserved Ejection Fraction (HFpEF) (based on invasive measurement) or high probability of HFpEF (>70% based on H2FPEF score ≥4)
* Ability to provide informed consent (knowledge of project languages), >18 years

Exclusion Criteria:

* MRI incompatibility (ie. pacemakers, ICD, internal defibrillators)
* Acute myocardial infarction (<90 days)
* Recent cardiovascular surgery or intervention (<90 days)
* Severe valve disease
* Known infiltrative diseases (i.e. amyloidosis, sarcoidosis)
* Known hypertrophic cardiomyopathy)
* ARVC (arrhythmogenic right ventricular cardiomyopathy), non-compaction cardiomyopathy
* Heart transplant
* Treatment for chemotherapy or radiotherapy
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible patients with heart failure and preserved ejection fraction (HFpEF) that agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiovascular events (MACE) | Within 5 years
  Composite outcome = the first occurrence of hospitalization for heart failure or all-cause mortality.

SECONDARY OUTCOMES:
Incidence of adverse clinical events | Within 5 years
  Incidence of the total adverse clinical events during the follow up time. Adverse clinical events are defined as the occurrence of: hospitalization for heart failure after the CMR, ICD implantation, sustained ventricular tachycardia, cardiac and non-cardiac death, revascularization therapy, valve repair/replacement, myocardial infarction, stroke, hospitalization for angina.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Gräni, PD Dr. PhD, Principal Investigator — Insel Gruppe AG, Inselspital, Universitätsklinik für Kardiologie; Kady Fischer, PhD, Principal Investigator — Insel Gruppe AG, Inselspital, Dept. Anaesthesiology and Pain Medicine
Locations (1):
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pieske B, Tschope C, de Boer RA, Fraser AG, Anker SD, Donal E, Edelmann F, Fu M, Guazzi M, Lam CSP, Lancellotti P, Melenovsky V, Morris DA, Nagel E, Pieske-Kraigher E, Ponikowski P, Solomon SD, Vasan RS, Rutten FH, Voors AA, Ruschitzka F, Paulus WJ, Seferovic P, Filippatos G. How to diagnose heart failure with preserved ejection fraction: the HFA-PEFF diagnostic algorithm: a consensus recommendation from the Heart Failure Association (HFA) of the European Society of Cardiology (ESC). Eur Heart J. 2019 Oct 21;40(40):3297-3317. doi: 10.1093/eurheartj/ehz641. PMID 31504452
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Rich JD, Burns J, Freed BH, Maurer MS, Burkhoff D, Shah SJ. Meta-Analysis Global Group in Chronic (MAGGIC) Heart Failure Risk Score: Validation of a Simple Tool for the Prediction of Morbidity and Mortality in Heart Failure With Preserved Ejection Fraction. J Am Heart Assoc. 2018 Oct 16;7(20):e009594. doi: 10.1161/JAHA.118.009594. PMID 30371285
- [Background] Taqueti VR, Solomon SD, Shah AM, Desai AS, Groarke JD, Osborne MT, Hainer J, Bibbo CF, Dorbala S, Blankstein R, Di Carli MF. Coronary microvascular dysfunction and future risk of heart failure with preserved ejection fraction. Eur Heart J. 2018 Mar 7;39(10):840-849. doi: 10.1093/eurheartj/ehx721. PMID 29293969
- [Background] Borlaug BA, Paulus WJ. Heart failure with preserved ejection fraction: pathophysiology, diagnosis, and treatment. Eur Heart J. 2011 Mar;32(6):670-9. doi: 10.1093/eurheartj/ehq426. Epub 2010 Dec 7. PMID 21138935
- [Background] Shah SJ, Lam CSP, Svedlund S, Saraste A, Hage C, Tan RS, Beussink-Nelson L, Ljung Faxen U, Fermer ML, Broberg MA, Gan LM, Lund LH. Prevalence and correlates of coronary microvascular dysfunction in heart failure with preserved ejection fraction: PROMIS-HFpEF. Eur Heart J. 2018 Oct 1;39(37):3439-3450. doi: 10.1093/eurheartj/ehy531. PMID 30165580
- [Background] Meijers WC, van der Velde AR, de Boer RA. Biomarkers in heart failure with preserved ejection fraction. Neth Heart J. 2016 Apr;24(4):252-8. doi: 10.1007/s12471-016-0817-7. PMID 26942916
- [Background] Jhund PS, Anand IS, Komajda M, Claggett BL, McKelvie RS, Zile MR, Carson PE, McMurray JJ. Changes in N-terminal pro-B-type natriuretic peptide levels and outcomes in heart failure with preserved ejection fraction: an analysis of the I-Preserve study. Eur J Heart Fail. 2015 Aug;17(8):809-17. doi: 10.1002/ejhf.274. Epub 2015 Apr 29. PMID 25921853
- [Background] Reddy YNV, Carter RE, Obokata M, Redfield MM, Borlaug BA. A Simple, Evidence-Based Approach to Help Guide Diagnosis of Heart Failure With Preserved Ejection Fraction. Circulation. 2018 Aug 28;138(9):861-870. doi: 10.1161/CIRCULATIONAHA.118.034646. PMID 29792299
- [Background] Nadruz W Jr, West E, Sengelov M, Santos M, Groarke JD, Forman DE, Claggett B, Skali H, Shah AM. Prognostic Value of Cardiopulmonary Exercise Testing in Heart Failure With Reduced, Midrange, and Preserved Ejection Fraction. J Am Heart Assoc. 2017 Oct 31;6(11):e006000. doi: 10.1161/JAHA.117.006000. PMID 29089342
- [Background] Schelbert EB, Fridman Y, Wong TC, Abu Daya H, Piehler KM, Kadakkal A, Miller CA, Ugander M, Maanja M, Kellman P, Shah DJ, Abebe KZ, Simon MA, Quarta G, Senni M, Butler J, Diez J, Redfield MM, Gheorghiade M. Temporal Relation Between Myocardial Fibrosis and Heart Failure With Preserved Ejection Fraction: Association With Baseline Disease Severity and Subsequent Outcome. JAMA Cardiol. 2017 Sep 1;2(9):995-1006. doi: 10.1001/jamacardio.2017.2511. PMID 28768311
- [Background] Fischer K, Yamaji K, Luescher S, Ueki Y, Jung B, von Tengg-Kobligk H, Windecker S, Friedrich MG, Eberle B, Guensch DP. Feasibility of cardiovascular magnetic resonance to detect oxygenation deficits in patients with multi-vessel coronary artery disease triggered by breathing maneuvers. J Cardiovasc Magn Reson. 2018 May 7;20(1):31. doi: 10.1186/s12968-018-0446-y. PMID 29730991
- [Background] Seemann F, Arvidsson P, Nordlund D, Kopic S, Carlsson M, Arheden H, Heiberg E. Noninvasive Quantification of Pressure-Volume Loops From Brachial Pressure and Cardiovascular Magnetic Resonance. Circ Cardiovasc Imaging. 2019 Dec;12(1):e008493. doi: 10.1161/CIRCIMAGING.118.008493. PMID 30630347
- [Background] Fischer K, Obrist SJ, Erne SA, Stark AW, Marggraf M, Kaneko K, Guensch DP, Huber AT, Greulich S, Aghayev A, Steigner M, Blankstein R, Kwong RY, Grani C. Feature Tracking Myocardial Strain Incrementally Improves Prognostication in Myocarditis Beyond Traditional CMR Imaging Features. JACC Cardiovasc Imaging. 2020 Sep;13(9):1891-1901. doi: 10.1016/j.jcmg.2020.04.025. Epub 2020 Jul 15. PMID 32682718
- [Background] Stoll VM, Hess AT, Rodgers CT, Bissell MM, Dyverfeldt P, Ebbers T, Myerson SG, Carlhall CJ, Neubauer S. Left Ventricular Flow Analysis. Circ Cardiovasc Imaging. 2019 May;12(5):e008130. doi: 10.1161/CIRCIMAGING.118.008130. PMID 31109184
- [Background] Karagodin I, Aba-Omer O, Sparapani R, Strande JL. Aortic stiffening precedes onset of heart failure with preserved ejection fraction in patients with asymptomatic diastolic dysfunction. BMC Cardiovasc Disord. 2017 Feb 14;17(1):62. doi: 10.1186/s12872-017-0490-9. PMID 28196483
- [Background] Jung B, Stalder AF, Bauer S, Markl M. On the undersampling strategies to accelerate time-resolved 3D imaging using k-t-GRAPPA. Magn Reson Med. 2011 Oct;66(4):966-75. doi: 10.1002/mrm.22875. Epub 2011 Mar 24. PMID 21437975
- [Background] Jung B, Muller C, Buchenberg W, Ith M, Reineke D, Beyersdorf F, Benk C. Investigation of hemodynamics in an in vitro system simulating left ventricular support through the right subclavian artery using 4-dimensional flow magnetic resonance imaging. J Thorac Cardiovasc Surg. 2015 Jul;150(1):200-7. doi: 10.1016/j.jtcvs.2015.02.048. Epub 2015 Feb 28. PMID 25840754
- [Background] Obmann VC, Marx C, Berzigotti A, Mertineit N, Hrycyk J, Grani C, Ebner L, Ith M, Heverhagen JT, Christe A, Huber AT. Liver MRI susceptibility-weighted imaging (SWI) compared to T2* mapping in the presence of steatosis and fibrosis. Eur J Radiol. 2019 Sep;118:66-74. doi: 10.1016/j.ejrad.2019.07.001. Epub 2019 Jul 2. PMID 31439261
- [Background] Ostovaneh MR, Ambale-Venkatesh B, Fuji T, Bakhshi H, Shah R, Murthy VL, Tracy RP, Guallar E, Wu CO, Bluemke DA, Lima JAC. Association of Liver Fibrosis With Cardiovascular Diseases in the General Population: The Multi-Ethnic Study of Atherosclerosis (MESA). Circ Cardiovasc Imaging. 2018 Mar;11(3):e007241. doi: 10.1161/CIRCIMAGING.117.007241. PMID 29523555
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Background] Shah KS, Xu H, Matsouaka RA, Bhatt DL, Heidenreich PA, Hernandez AF, Devore AD, Yancy CW, Fonarow GC. Heart Failure With Preserved, Borderline, and Reduced Ejection Fraction: 5-Year Outcomes. J Am Coll Cardiol. 2017 Nov 14;70(20):2476-2486. doi: 10.1016/j.jacc.2017.08.074. Epub 2017 Nov 12. PMID 29141781
- [Background] Roy C, Slimani A, de Meester C, Amzulescu M, Pasquet A, Vancraeynest D, Vanoverschelde JL, Pouleur AC, Gerber BL. Age and sex corrected normal reference values of T1, T2 T2* and ECV in healthy subjects at 3T CMR. J Cardiovasc Magn Reson. 2017 Sep 21;19(1):72. doi: 10.1186/s12968-017-0371-5. PMID 28934962
- [Background] Kramer CM, Barkhausen J, Flamm SD, Kim RJ, Nagel E; Society for Cardiovascular Magnetic Resonance Board of Trustees Task Force on Standardized Protocols. Standardized cardiovascular magnetic resonance (CMR) protocols 2013 update. J Cardiovasc Magn Reson. 2013 Oct 8;15(1):91. doi: 10.1186/1532-429X-15-91. PMID 24103764
- [Background] Turkbey EB, Nacif MS, Guo M, McClelland RL, Teixeira PB, Bild DE, Barr RG, Shea S, Post W, Burke G, Budoff MJ, Folsom AR, Liu CY, Lima JA, Bluemke DA. Prevalence and Correlates of Myocardial Scar in a US Cohort. JAMA. 2015 Nov 10;314(18):1945-54. doi: 10.1001/jama.2015.14849. PMID 26547466
- [Background] Bruder O, Schneider S, Nothnagel D, Pilz G, Lombardi M, Sinha A, Wagner A, Dill T, Frank H, van Rossum A, Schwitter J, Nagel E, Senges J, Sabin G, Sechtem U, Mahrholdt H. Acute adverse reactions to gadolinium-based contrast agents in CMR: multicenter experience with 17,767 patients from the EuroCMR Registry. JACC Cardiovasc Imaging. 2011 Nov;4(11):1171-6. doi: 10.1016/j.jcmg.2011.06.019. PMID 22093267
- See also: Ordinance on Human Research with the Exception of Clinical trials (HRO) — https://www.admin.ch/opc/en/classified-compilation/20121177/index.html
- See also: Human Research Act (HRA) — http://www.admin.ch/opc/en/classified-compilation/20121176/201401010000/810.305.pdf
- See also: Declaration of Helsinki — https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects
- See also: STROBE statement — http://www.jclinepi.com/article/S0895-4356(07)00436-2/pdf
- See also: P429 Combining systolic and diastolic feature tracking myocardial strain parameters for a more comprehensive assessment of the different characteristics in HFpEF — https://esc365.escardio.org/Congress/EuroCMR-2019/Poster-session-2/191780-combining-systolic-and-diastolic-feature-tracking-myocardial-strain-parameters-for-a-more-comprehensive-assessment-of-the-different-characteristics-in-hfpef